CLINICAL TRIAL: NCT00968461
Title: A Phase I Study of Phenethyl Isothiocyanate (PEITC) in Patients With Lymphoproliferative Disorders Previously Treated With Fludarabine
Brief Title: Study of Phenethyl Isothiocyanate in Lymphoproliferative Disorders
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0622
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Lymphoproliferative Disorders
Keywords: Chronic lymphocytic leukemia; CLL; PEITC; Phenethyl Isothiocyanate; Fludarabine
MeSH Terms: conditions — Leukemia; Lymphoproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — phenethyl isothiocyanate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phenethyl Isothiocyanate (PEITC) (Experimental): Starting dose 40 mg capsules by mouth, 4 times a day, on Days 1-3 and 8-10 of each cycle.
  Interventions: Drug: Phenethyl Isothiocyanate (PEITC)

INTERVENTIONS:
Drug: Phenethyl Isothiocyanate (PEITC) — Starting dose 40 mg capsules by mouth, 4 times a day, on Days 1-3 and 8-10 of each cycle.

SUMMARY:
The goal of this clinical research study is to learn the highest tolerable dose of phenethyl isothiocyanate (PEITC) that can be given to patients who have a lymphoproliferative disorder that has been treated with fludarabine. The safety of PEITC will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

PEITC is designed to cause build-up of specific molecules in cells, which may damage cancer cells and cause the cells to die.

Study Drug Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of PEITC based on when you joined this study. Up to 9 dose levels of PEITC will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of PEITC is found.

Study Drug Administration:

Every 28 days in this study is 1 "cycle." You will take PEITC capsules by mouth, 4 times a day, on Days 1-3 and 8-10 of each cycle. You should take each dose with a cup (8 ounces) of water, either with or without food. The doses should be taken at the same times each day (about 7:00 AM, 12 noon, 5:00 PM, and 10:00 PM).

Study Visits:

Once a week, blood (about 1 tablespoon each time) will be drawn for routine tests. These weekly blood draws will occur on Days 1, 8, 15, and 21 of each cycle, +/- 3 days.

Follow-up After Completion of Cycle 3:

Four (4) weeks after the start of the third cycle, the following tests and procedures will be performed:

* You will have a complete physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspiration, fine-needle aspiration (FNA), and/or biopsy in order to check the status of the disease.

PK and PD Testing:

This study involves blood draws for pharmacokinetic (PK) and pharmacodynamic (PD) testing. PK testing measures the amount of study drug in the body at different time points. PD testing is used to look at how the level of study drug in your body may affect the disease.

Blood (about 1 tablespoon each time) will be drawn and used for both of these tests, on the following schedule:

* Day 1 of Cycle 1 (or possibly the day before Day 1)
* Days 1, 2, and 3 of Cycle 1 (at 4 hours after that day's first dose of PEITC)
* Day 4 of Cycle 1 (at 12 hours after your last dose of PEITC)

Length of Study Participation:

You may receive up to 6 cycles (24 weeks) of the study drug. You will be taken off the study drug early if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

At the end of your last study cycle, you will have a complete physical exam, including measurement of your vital signs.

In addition, unless the disease has completely responded, the following tests and procedures will be performed at the end-of-study visit:

* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspiration and/or biopsy to check the status of the disease, if the study doctor thinks it is necessary.

Follow-Up Visits:

Every 3 to 6 months after the end of your last study cycle, you will have a bone marrow aspiration and/or biopsy if the study doctor thinks it is necessary to check the status of the disease in this way.

Every 3 to 6 months after the end of your last study cycle, you will have a complete physical exam, including measurement of vital signs.

After the follow-up visit at 24 weeks after the end of your last study cycle, the schedule of your follow-up physical exams will be every 3 to 6 months. These visits may include a blood draw and bone marrow aspiration. Your study doctor will decide if these tests are needed. If the disease returns during this time, however, you will be considered off-study. This means you will also no longer have the follow-up bone marrow samples collected as part of this study.

This is an investigational study. PEITC is not commercially available or FDA approved. At this time, it is only being used in research.

Up to 54 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a histologically or cytologically confirmed lymphoproliferative disorder previously treated with fludarabine are eligible for this protocol.
2. Patients must be 18 years of age or older.
3. Patients must have a performance status of 0-2 (Zubrod scale).
4. Patients must have adequate renal function (serum creatinine </= 2 mg/dL or creatinine clearance > 50 mL/min). Patients with renal dysfunction due to organ infiltration by disease may be eligible after discussion with the P.I. and consideration of appropriate dose adjustments.
5. Patients must have adequate function (bilirubin </= 2.0 mg/dl; SGOT or SGPT </= 3X the ULN for the reference lab unless due to leukemia or congenital hemolytic disorder [for bilirubin]). Patients with hepatic dysfunction due to organ infiltration by disease may be eligible after discussion with the P.I. and consideration of appropriate dose adjustments.
6. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

1. Untreated or uncontrolled life-threatening infection (Grade 4 infection, i.e. septic shock, hypotension, acidosis, necrosis).
2. Pregnancy or breastfeeding. Female patients of childbearing potential (including those <1 year postmenopausal) and male patients must agree to use contraception. A female of child bearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
3. Chemotherapy and/or radiation therapy within 4 weeks of study enrollment.
4. Any other medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to give informed consent or cooperate and participate in the study or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Day Cycle

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org